CLINICAL TRIAL: NCT03193814
Title: Study Evaluating the Safety and Efficacy of FOLFOX Plus Apatinib or FOLFIRI Plus Apatinib as Second-line Therapy in Metastatic Colorectal Cancer
Brief Title: Safety and Efficacy Study of Chemotherapy Plus Apatinib as Second-line Therapy in Metastatic Colorectal Cancer
Acronym: XHZL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate patient enrollment
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Tao Zhang, Chief of Gastrointestinal Oncology Department, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XHZL
Record Dates: First submitted 2017-06-17; First posted 2017-06-21 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Colorectal Cancer; Chemotherapy; Angiogenesis
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Therapy; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy + Apatinib (Experimental): chemotherapy regimens include: Folfox (Oxaplatin 85 mg/m2 IV over 2 hours, day 1; Leucovorin 400 mg/m2 over 2 hours, day 1; 5-FU 400 mg/m2 IV bolus on day 1, then 1200mg/m2/day x 2 days; repeat every 2 weeks) or Folfiri (Irinotecan 150-180 mg/m2 IV over 30-90 minutes, day 1; Leucovorin 400 mg/m2 over 2 hours, day 1; 5-FU 400 mg/m2 IV bolus on day 1, then 1200mg/m2/day x 2 days; repeat every 2 weeks)； apatinib 500mg po qd
  Interventions: Drug: Chemotherapy + Apatinib

INTERVENTIONS:
Drug: Chemotherapy + Apatinib — chemotherapy regimens could be folfox or folfiri; apatinib 500mg po qd
  Other Names: chemotherpy plus apatinib mesylate

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of apatinib in combination with second-line FOLFOX or FOLFIRI for metastatic colorectal cancer in patients with disease progression during or after first-line therapy.

DETAILED DESCRIPTION:
Angiogenesis is an important therapeutic target in metastatic colorectal carcinoma. Apatinib is a potent oral inhibitor of the intracellular domain and emerging as original antiangiogenic opportunities. We assessed the efficacy and safety of apatinib in combination with second-line FOLFOX or FOLFIRI for metastatic colorectal cancer in patients with disease progression during or after first-line therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed inoperable colorectal adenocarcinoma excluding vermiform appendix cancer and anal canal cancer
2. Age ≥18 years at the time of informed consent
3. ECOG performance status (PS) of 0-1
4. Written informed consent prior to study-specific screening procedures
5. Life expectancy of at least 90 days
6. Withdrawal from first-line chemotherapy (regardless of containing molecular-targeted drugs) for metastatic colorectal cancer due to intolerable toxicity or progressive disease, or relapse within 180 days after the last dose of adjuvant chemotherapy
7. Adequate organ function according to following laboratory values obtained within 14 days before enrolment (excluding patients who received blood transfusions or hematopoietic growth factors within 14 days before the laboratory test) Neutrophil count: ≥1500/mm3 Platelet count: ≥10.0 x 104/mm3 Hemoglobin: ≥9.0 g/dL Total bilirubin: ≤1.5 mg/dL AST, ALT: ≤100 IU/L (≤200 IU/I if liver metastases present) Serum creatinine: ≤1.5 mg/dL
8. Measurable or nonmeasurable disease based on the Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1)
9. Adequate coagulation function [International Normalized Ratio (INR) ≤1.5 and Partial Thromboplastin Time (PTT) or activated PTT (aPTT) ≤1.5 x upper limit of normal (ULN)). Participants on full-dose anticoagulation must be on a stable dose of anticoagulant therapy and if on oral anticoagulation, must have an INR ≤3 and have no clinically significant active bleeding or pathological condition that carries a high risk of bleeding
10. Consent to provide a historical colorectal cancer tissue sample for assessment of biomarkers and the tumor tissue sample is available
11. Ability to provide signed informed consent

Exclusion Criteria:

1. History of other malignancy with a disease-free interval <5 years (other than curatively treated cutaneous basal cell carcinoma, curatively treated carcinoma in situ of the cervix, and gastroenterological cancer confirmed to be cured by endoscopic mucosal resection)
2. With massive pleural effusion or ascites requiring intervention
3. Radiological evidence of brain tumor or brain metastases
4. Active infection including hepatitis
5. Any of the following complication: i) Gastrointestinal bleeding or gastrointestinal obstruction (including paralytic ileus) ii) Symptomatic heart disease (including unstable angina, myocardial infarction, and heart failure) iii) Interstitial pneumonia or pulmonary fibrosis iv) Uncontrolled diabetes mellitus v) Uncontrolled diarrhea (that interferes with daily activities despite adequate therapy)
6. Any of the following medical history: Myocardial infarction: History of one episode within one year before enrollment or two or more lifetime episodes i) Serious hypersensitivity to any of the study drugs ii) History of adverse reaction to fluoropyrimidines suggesting dihydropyrimidine dehydrogenase (DPD) deficiency
7. Pregnant or lactating females, and males and females unwilling to use contraception
8. Psychiatric disability that would preclude study compliance
9. Otherwise determined by the investigator to be unsuitable for participation in the study
10. Concurrent gastrointestinal perforation or history of gastrointestinal perforation with 1 year before enrollment
11. History of pulmonary hemorrhage/hemoptysis ≥ Grade 2 (defined as bright red blood of at least 2.5mL) within 1 month prior to enrollment.
12. History of laparotomy, thoracotomy, or intestinal resection within 28 days before enrollment
13. Unhealed wound (except suture wounds from implantation of a central venous port), gastrointestinal ulcer, or traumatic fracture
14. Current or recent (within 1 year) thromboembolism or cerebrovascular disease
15. Currently receiving or requires anticoagulation therapy (> 325 mg/day of aspirin)
16. Bleeding diathesis, coagulopathy, or coagulation factor abnormality (INR ≥1.5 within 14 days before enrollment)
17. Uncontrolled hypertension
18. Urine dipstick for proteinuria >+2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) Time | 2 years
  PFS was defined as the time from the date of randomization until the date of objectively determined progressive disease (PD) [according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v). 1.1] or death due to any cause, whichever was first. PD is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm). Participants who died without a reported prior progression were considered to have progressed on the day of their death. Participants who did not progress or were lost to follow-up were censored at the day of their last radiographic tumor assessment.

SECONDARY OUTCOMES:
Percentage of Participants Achieving an Objective Response (Objective Response Rate) | 1 year
  The objective response rate is equal to the proportion of participants achieving a best overall response of partial response or complete response (PR + CR). Response was defined using RECIST, v. 1.1 criteria. CR was defined as the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm and normalization of tumor marker level of non-target lesions; PR was defined as having at least a 30% decrease in sum of longest diameter of target lesions taking as reference the baseline sum diameter.
Overall Survival (OS) | 2 years
  OS was defined as the time in months from the date of randomization to the date of death from any cause. For participants not known to have died as of the cut-off date, OS was censored at the last known date alive.

REFERENCES:
- [Background] Tabernero J, Yoshino T, Cohn AL, Obermannova R, Bodoky G, Garcia-Carbonero R, Ciuleanu TE, Portnoy DC, Van Cutsem E, Grothey A, Prausova J, Garcia-Alfonso P, Yamazaki K, Clingan PR, Lonardi S, Kim TW, Simms L, Chang SC, Nasroulah F; RAISE Study Investigators. Ramucirumab versus placebo in combination with second-line FOLFIRI in patients with metastatic colorectal carcinoma that progressed during or after first-line therapy with bevacizumab, oxaliplatin, and a fluoropyrimidine (RAISE): a randomised, double-blind, multicentre, phase 3 study. Lancet Oncol. 2015 May;16(5):499-508. doi: 10.1016/S1470-2045(15)70127-0. Epub 2015 Apr 12. PMID 25877855
- [Background] Li J, Qin S, Xu J, Xiong J, Wu C, Bai Y, Liu W, Tong J, Liu Y, Xu R, Wang Z, Wang Q, Ouyang X, Yang Y, Ba Y, Liang J, Lin X, Luo D, Zheng R, Wang X, Sun G, Wang L, Zheng L, Guo H, Wu J, Xu N, Yang J, Zhang H, Cheng Y, Wang N, Chen L, Fan Z, Sun P, Yu H. Randomized, Double-Blind, Placebo-Controlled Phase III Trial of Apatinib in Patients With Chemotherapy-Refractory Advanced or Metastatic Adenocarcinoma of the Stomach or Gastroesophageal Junction. J Clin Oncol. 2016 May 1;34(13):1448-54. doi: 10.1200/JCO.2015.63.5995. Epub 2016 Feb 16. PMID 26884585